CLINICAL TRIAL: NCT03241940
Title: Phase I Dose Escalation Study of CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: Study of CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults w/ Recurrent or Refractory B Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-41383; NCI-2017-01415 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PEDSCCT5007 (Other: Stanford Cancer Institute); IRB-41383 (Other: Stanford IRB)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: B Acute Lymphoblastic Leukemia; CD19 Positive; Minimal Residual Disease; Philadelphia Chromosome Positive; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Neoplasm, Residual; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive; Cyclophosphamide; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD19/CD22-CAR T cells, chemotherapy) (Experimental): Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and cyclophosphamide IV over 60 minutes on day -2. Patients then receive CD19/CD22-CAR T cells IV over 10-20 minutes on day 0. Patients that benefited from the first dose of CD19/CD22-CAR T cells, had no unacceptable side effects, and have enough cells left over may receive 2 or 3 additional doses of CD19/CD22-CAR T cells.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given CD19/CD22-CAR T cells IV
  Other Names: CAR T-cell therapy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the best dose and side effects of CD19/CD22 chimeric antigen receptor (CAR) T cells when given together with chemotherapy, and to see how well they work in treating children or young adults with CD19 positive B acute lymphoblastic leukemia that has come back or does not respond to treatment. A CAR is a genetically-engineered receptor made so that immune cells (T cells) can attack cancer cells by recognizing and responding to the CD19/CD22 proteins. These proteins are commonly found on B acute lymphoblastic leukemia. Drugs used in chemotherapy, such as fludarabine phosphate and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CD19/CD22-CAR T cells and chemotherapy may work better in treating children or young adults with B acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility of producing CD19/CD22-CAR T cells meeting the established release criteria.

II.Assess the safety of administering escalating doses of autologous CD19/CD22-CAR T cells that meet established release specifications in children and young adults with B-cell hematologic malignancies following a cyclophosphamide/fludarabine conditioning regimen. The following dose escalation will be used in two disease groups: 1) children and young adults with relapsed/refractory low disease burden ALL (< 5% blasts), and 2) children and young adults with relapsed/refractory high disease burden ALL (≥5% blasts) or lymphoma:

1. Dose Level -1: 3 x 105 transduced T cells/kg (± 20%)
2. Dose Level 1: 1 x 106 transduced T cells/kg (± 20%)
3. Dose Level 2: 3 x 106 transduced T cells/kg (± 20%)
4. Dose Level 3: 1 x 107 transduced T cells/kg (± 20%)

SECONDARY OBJECTIVES:

I. Evaluate the ability of CD19/CD22-CAR T cells to mediate clinical activity in children and young adults with B-acute lymphoblastic leukemia (ALL).

TERTIARY OBJECTIVES:

I. Analyze alterations in early B cell development induced by immune pressure exerted via CD19/CD22-CAR T cells.

II. Evaluate whether subjects receiving CD19/CD22-CAR T cells relapse with loss or diminished expression of CD19 and/or CD22, when feasible.

III. Measure persistence of CD19/CD22-CAR T cells in the blood, bone marrow and cerebral spinal fluid (CSF), and explore correlations between CD19/CD22-CAR T cell properties and CAR T cell efficacy and persistence.

IV. Establish the utility of chromatin structure and epigenomic technology to characterize CAR T cell therapies.

V. Explore the ability of CD19/CD22-CAR T cells to mediate clinical activity in children and young adults with refractory B cell lymphoma in a non-statistical cohort due to expectations of low accrual.

OUTLINE: This is a dose-escalation study of CD19/CD22-CAR T cells.

Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -4 to -2 and cyclophosphamide IV over 60 minutes on day -2. Patients then receive CD19/CD22-CAR T cells IV over 10-20 minutes on day 0. Patients that benefited from the first dose of CD19/CD22-CAR T cells, had no unacceptable side effects, and have enough cells left over may receive 2 or 3 additional doses of CD19/CD22-CAR T cells.

After completion of study treatment, patients are followed up daily until day 14, twice weekly until day 28, at 2 and 3 months, every 3 months until month 12, every 6-12 months up to year 5, and then annually for years 6-15.

ELIGIBILITY:
1.1 INCLUSION CRITERIA

1. Diagnosis: ALL In view of the PI and the primary oncologist, there must be no available alternative curative therapies or subject has declined to pursue alternative therapy; and subjects must be either ineligible for allogeneic stem cell transplant (SCT), have refused SCT, recurred after SCT, or have disease activity that prohibits SCT at the time of enrollment.

   1. Chemotherapy refractory disease in subjects with B-ALL is defined as progression or stable disease after two lines of therapies
   2. Recurrence of disease after achieving a complete response (CR).
   3. Subjects with persistent or relapsed minimal residual disease (MRD) (by flow cytometry, PCR, FISH, or next generation sequencing) require verification of MRD positivity on two occasions at least 4 weeks apart.
   4. Subjects with Philadelphia Chromosome positive acute lymphoblastic leukemia (Ph+ALL) subjects are eligible if they progressed, had stable disease or relapsed after two lines of therapy, including tyrosine kinase inhibitors (TKIs).
   5. Subjects with recurrence of isolated CNS relapse after achieving complete remission (CR); if relapsed with MRD, will require verification of MRD positivity on two occasions at least 4 weeks apart.
2. Diagnosis: Lymphoma Subjects with lymphoma must have progressed, had SD, or recurred after initial treatment regimens that include an anthracycline and an anti CD20 monoclonal antibody. Subjects who relapse ≥12 months after therapy should have progressed after autologous transplant or been ineligible for autologous transplant.
3. CD19 expression CD19 expression is required at any time since diagnosis. If patient has received anti-CD19 targeted therapy (i.e. Blinatumomab), then CD19 expression must be subsequently demonstrated. CD19 expression. must be detected on greater than 50% of the malignant cells by immunohistochemistry or ≥ 90% by flow cytometry. The choice of whether to use flow cytometry or immunohistochemistry will be determined by what is the most easily available tissue sample in each subject. In general, immunohistochemistry will be used for lymph node biopsies, flow cytometry will be used for peripheral blood and bone marrow samples.
4. Subjects who have undergone autologous SCT with disease progression or relapse following SCT will be eligible if all other eligibility criteria are met. Subjects who have undergone allogeneic SCT will be eligible if, in addition to meeting other eligibility criteria, they are at least 100 days post-transplant, they have no evidence of active GVHD and have been without immunosuppressive agents for at least 30 days.
5. Subjects who have undergone prior anti-CD19 or anti-CD22 CAR therapy will be eligible if < 5% of circulating levels of CD3+ cells express the previous CAR by flow cytometry.
6. Must have evaluable or measurable disease; subjects with lymphoma must have evaluable or measurable disease according to the revised IWG Response Criteria for Malignant Lymphoma[66] must be present. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy.
7. At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives.

   Exceptions:

   f. There is no time restriction with regard to prior intrathecal chemotherapy (incl. steroids) provided there is complete recovery from any acute toxic effects of such; g. Subjects receiving hydroxyurea may be enrolled provided there has been no increase in dose for at least 2 weeks prior to starting apheresis; h. Subjects who are on standard ALL maintenance type chemotherapy (vincristine, 6-mercaptopurine or oral methotrexate) may be enrolled provided that chemotherapy is discontinued at least 1 week prior to apheresis.

   i. Subjects receiving steroid therapy at physiologic replacement doses (≤ 5 mg/day of prednisone or equivalent doses of other corticosteroids) only are allowed provided there has been no increase in dose for at least 2 weeks prior to starting apheresis; j. For radiation therapy: Radiation therapy must have been completed at least 3 weeks prior to enrollment, with the exception that there is no time restriction if the volume of bone marrow treated is less than 10% and also the subject has measurable/evaluable disease outside the radiation port.
8. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities, such as alopecia, nutritional support measures, electrolyte abnormalities, or those not impacting the investigator's ability to assess treatment emergent toxicities)
9. Age Greater than or equal to 1 year of age and less than or equal to 30 years of age at time of enrollment; must meet parameters for apheresis per institutional guidelines. NOTE: The first subject in the first dose cohort must be ≥ 18 years of age if an adult has not been treated at that dose cohort on the companion Stanford protocol "Phase 1 Dose Escalation Study of CD19/CD22 Chimeric Antigen Receptor (CAR) T Cells in Adults with Recurrent or Refractory B Cell Malignancies" and undergone safety evaluation at Day 28 without evidence of DLT.
10. Performance Status: Subjects > 10 years of age: Karnofsky ≥ 50%; Subjects ≤ 10 years of age: Lansky scale ≥ 50% (See Appendix B Section 14.2)
11. Normal Organ and Marrow Function (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion)

    1. ANC ≥750/uL*
    2. Platelet count ≥50,000/uL*
    3. Absolute lymphocyte count ≥150/uL*
    4. Adequate renal, hepatic, pulmonary and cardiac function defined as:

       * Serum ALT/AST ≤10 ULN (unless elevated ALT/AST is attributed to leukemia or lymphoma involvement of the liver, in which case this criterion will be waived and not disqualify a patient).
       * Total bilirubin ≤1.5 mg/dl, except in subjects with Gilbert's syndrome.
       * Cardiac ejection fraction ≥ 45%, no evidence of physiologically significant pericardial effusion as determined by an ECHO, and no clinically significant ECG findings
       * No clinically significant pleural effusion
       * Baseline oxygen saturation >92% on room air at rest
       * creatinine: within age adjusted normal institutional limits (see table below) OR
       * creatinine clearance ≥60 mL/min/1.73 m2 (as estimated by Cockcroft Gault Equation) for subjects with creatinine levels above institutional normal.

    Age (Years) Maximum Serum Creatinine (mg/dL)

    ≤5 0.8 5 < age ≤ 10 1.0 >10 1.2

    * if these cytopenias are not judged by the investigator to be due to underlying disease (i.e. potentially reversible with anti-neoplastic therapy); A subject will not be excluded because of pancytopenia ≥ Grade 3 if it is due to disease, based on the results of bone marrow studies.
12. CNS Status

    1. Subjects with ALL

       Subjects with the following CNS status are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy:
       * CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs;
       * CNS 2, defined as presence of < 5/µL WBCs in CSF and cytospin positive for blasts, or > 5/µL WBCs but negative by Steinherz/Bleyer algorithm:

         * CNS 2a: <10/µL RBCs; < 5/µL WBCs and cytospin positive for blasts;
         * CNS 2b: ≥10/µL RBCs; < 5/µL WBCs and cytospin positive for blasts;
         * CNS 2c: ≥10/µL RBCs; ≥5/µL WBCs and cytospin positive for blasts but negative by Steinherz/Bleyer algorithm.
    2. Subjects with lymphoma

    Subjects must have no signs or symptoms of CNS disease or detectable evidence of CNS disease on MRI at the time of screening. Subjects who have previously been treated for CNS disease and who have the following CNS status will be eligible:
    * CNS 1, defined as absence of blasts in cerebral spinal fluid (CSF) on cytospin preparation, regardless of the number of WBCs;
    * CNS 2, defined as presence of < 5/µL WBCs in CSF and cytospin positive for blasts, or > 5/µL WBCs but negative by Steinherz/Bleyer algorithm:

      * CNS 2a: < 10/µL RBCs; < 5/µL WBCs and cytospin positive for blasts;
      * CNS 2b: ≥ 10/µL RBCs; < 5/µL WBCs and cytospin positive for blasts;
      * CNS 2c: ≥ 10/µL RBCs; ≥ 5/µL WBCs and cytospin positive for blasts but negative by Steinherz/Bleyer algorithm.
13. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
14. Contraception Subjects of child-bearing or child-fathering potential must be willing to practice birth control from the time of enrollment on this study and for four (4) months after receiving the preparative regimen.

    Females of child-bearing potential must have a negative pregnancy test because of the potentially dangerous/unknown effects on the fetus.
15. Ability to give informed consent. All subjects ≥ 18 years of age must be able to give informed consent. For subjects <18 years old their legal authorized representative (LAR) (i.e. parent or guardian) must give informed consent. Pediatric subjects will be included in age appropriate discussion and verbal assent will be obtained for those > 7 years of age, when appropriate.

1.2 EXCLUSION CRITERIA

Subjects meeting any of the following criteria are not eligible for participation in the study:

1. Recurrent or refractory ALL limited to isolated testicular.
2. Subjects with radiologically-detected CNS lymphoma or CNS 3 disease (presence of ≥ 5/µL WBCs in CSF and cytospin positive for blasts [in the absence of a traumatic lumbar puncture] and/or clinical signs of CNS leukemia).
3. Hyperleukocytosis (≥ 50,000 blasts/µL) or rapidly progressive disease that in the estimation of the investigator and sponsor would compromise ability to complete study therapy.
4. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) unless disease free for at least 3 years.
5. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.

   Ongoing infection with HIV or hepatitis B (HBsAg positive) or hepatitis C virus (anti-HCV positive) as the immunosuppression contained in this study will pose unacceptable risk. A history of hepatitis B or hepatitis C is permitted if the viral load is undetectable per quantitative PCR and/or nucleic acid testing.
6. CNS disorder such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or autoimmune disease with CNS involvement that in the judgment of the investigator may impair the ability to evaluate neurotoxicity.
7. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment, or have cardiac atrial or cardiac ventricular lymphoma involvement.
8. Subjects receiving anticoagulation therapy.
9. Any medical condition that in the judgement of the principal investigator is likely to interfere with assessment of safety or efficacy of study treatment
10. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
11. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the conditioning lymphodepletion chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
12. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.
13. May not have primary immunodeficiency or history of systemic autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2035-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) following chemotherapy preparative regimen and infusion of CD19/CD22 chimeric antigen receptor (CAR) T cells | Up to 28 days
  Will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 at three dose levels until the maximum tolerated dose (MTD) is determined.
Rate of successful manufacture and expansion of the CD19/CD22 chimeric antigen receptor (CAR) T cells to satisfy the targeted dose level and meet the required release specifications outlined in the Certificate of Analysis (COA) | 10-14 days after apheresis or thawing of cryopreserved peripheral blood mononuclear cell
  The number of subjects which can successfully manufacture the targeted dose number will be determined for each dose cohort.

SECONDARY OUTCOMES:
The ability to achieve a clinical response after administration of CD19/CD22 chimeric antigen receptor (CAR) T cells | Up to 15 years
  Will be assessed by the Response Criteria for Lymphoma and the Response Criteria for Acute Lymphoblastic Leukemia.

OTHER OUTCOMES:
Alterations in early B cell development induced by immune pressure exerted via CD19/CD22-CAR T cells | Up to 15 years
  Will be analyzed.
CD19/CD22 chimeric antigen receptor (CAR) T cell properties | Up to 15 years
  Will explore correlations with CAR T cell efficacy and persistence.
Frequency of CD22+ expression on lymphoma cells | Up to 15 years
  Will determine site density when possible.
Persistence of CD19/CD22 chimeric antigen receptor (CAR) T cells blood, bone marrow, and cerebral spinal fluid (CSF) | Up to 15 years
  Will be measured.
Relapse with loss or diminished expression of CD19 and/or CD22 | Up to 15 years
  Will be evaluated when feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Mackall, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh N. Modified T cells as therapeutic agents. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):296-302. doi: 10.1182/hematology.2021000262. PMID 34889384
- [Derived] Schultz L, Patel S, Davis KL, Ramakrishna S, Sahaf B, Bhatia N, Baggott C, Erickson C, Majzner RG, Oak J, Bertaina A, Mackall C, Feldman S. Identification of dual positive CD19+/CD3+ T cells in a leukapheresis product undergoing CAR transduction: a case report. J Immunother Cancer. 2020 Sep;8(2):e001073. doi: 10.1136/jitc-2020-001073. PMID 32929049